CLINICAL TRIAL: NCT00555464
Title: A Phase II, Randomized, Clinical Trial Assessing Efficacy And Safety Of Oral Prednisolone vs Intravenous Vincristine In The Treatment Of Infantile
Brief Title: Clinical Trial of Vincristine vs. Prednisolone for Treatment of Complicated Hemangiomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The introduction of oral propranolol as a highly efficacious agent for infantile hemangiomas
Sponsor: Medical College of Wisconsin (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beth Drolet, Professor of Dermatology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3429; #FDA-R-003429-01
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Hemangioma
Keywords: hemangioma, steroid, prednisolone, vincristine
MeSH Terms: conditions — Hemangioma | interventions — Vincristine; Prednisone; Solutions; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vincristine is a drug that has been used to treat cancers in children (including infants). It has been effective in treating a small number of infants with hemangiomas, most of whom failed previous therapies including steroids. Vincristine must be administered into a vein. Given the encouraging response data and documented safety record, Vincristine is a good choice for a clinical trial treating infants with complicated hemangiomas.
  Interventions: Drug: Vincristine
- 2 (Active Comparator): The standard treatment for hemangioma at most centers is oral steroids (Prednisolone). Prednisolone has been used to stop the growth of infantile hemangiomas that are life threatening, that could harm important functions, or are likely to result in severe disfigurement (scarring) without treatment.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Vincristine — Vincristine (0.05 mg/kg/dose) will be administered into a vein (PICC line) every week for 12 weeks. If assigned to receive Vincristine, a PICC line will be placed by a doctor who is a specialist in this procedure, an interventional radiologist. This will require sedation and when possible, will be coordinated with sedation for the MRI.
  Other Names: VINCRISTINE SULFATE (Oncovin®, VCR, LCR) NSC #67574 (042006)
  Arms: 1
Drug: Prednisone — Prednisolone given at 3 mg/kg/day by mouth for 12 week
  Other Names: PREDNISOLONE SODIUM PHOSPHATE SYRUP/SOLUTION 15mg/5 cc (Orapred®)
  Arms: 2

SUMMARY:
The goal of this study is to determine the safety and efficacy of Prednisolone and Vincristine for treatment of large, complicated infantile hemangiomas. The diagnostic, therapeutic and response criteria experimentally determined in this study will be used as a framework for future infantile hemangioma studies.

DETAILED DESCRIPTION:
Infants with large hemangiomas are often treated systemically with oral steroids (Prednisolone) to prevent complications. The best treatment for hemangiomas is not known and there are no medications approved by the FDA for treatment of hemangiomas. Also, the best method to measure the response of hemangioma to treatment is not known. Patients enrolling on this study will be randomly assigned to receive either daily Prednisolone by mouth or weekly Vincristine in a vein. Response to treatment will be monitored by clinical exams every two weeks and by an MRI at study entry and six and twelve weeks later. Patients with evidence of progressive disease (larger hemangiomas) on the week 6 MRI will be switched to the other drug to complete a total of 12 weeks of therapy. Side effects of each medication will be monitored closely determined from histories, physical exams, blood tests and other studies as necessary. Participation in this study will last up to 12 weeks and follow up for protocol.

ELIGIBILITY:
Inclusion Criteria:

* Children age 0-6 months old.
* Infants with infantile hemangiomas with complications that require systemic therapy to control their growth. To be eligible for enrollment infants must have clear indications for systemic treatment.
* Clinical diagnosis of infantile hemangioma confirmed by tissue biopsy positive for GLUT-1 Immunohistochemical staining. If the risk of bleeding or permanent disfigurement from biopsy is believed to be too great then clinical and radiological characteristics may be used to establish the diagnosis after discussion with the study PI. Patients with GLUT-1 negative vascular tumors such as Kaposiform hemangioendothelioma, tufted angioma, and angiosarcoma are not eligible.
* Hemangiomas must be greater than or equal to 50 cm2 clinically measured by taking the product of the two largest perpendicular diameters and have one of the following complications: ulceration, impairment of vision, impairment of hearing, obstruction of the airway, high output cardiac failure, bleeding, abdominal distention and/or compartment syndrome, compression of the spinal cord, or high risk of permanent disfigurement.
* Adequate liver function defined as:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age, and
  * SGPT(serum glutamate pyruvate transaminase) (ALT) < 2.5 x upper limit of normal (ULN) for age.
* Patients who have received topical or intralesional corticosteroids are eligible to be enrolled. A washout of one week is required prior to study enrollment. Patients who have undergone surgical resection are eligible if they meet all inclusion criteria after surgery.
* All patients' parents or legal guardians must sign a written informed consent. All institutional and FDA requirements for human studies must be met.

Exclusion Criteria:

* Children greater then 6 months old.
* Contraindications to Vincristine: previously diagnosed neuropathy including sensory neuropathy type 1, Charcot- Marie-Tooth or childhood poliomyelitis.
* Hemangioma involving the central nervous system (CNS) as Vincristine has poor CNS penetration.
* Infants who have received prior systemic therapy with corticosteroids (oral or intravenous), interferon or Vincristine are not eligible for enrollment.
* Patients receiving Vincristine who concomitantly require oral steroids for treatment of non-hemangioma indications such as asthma or atopic dermatitis will be removed from study.
* A life-threatening intercurrent infection.
* Infants with an underlying illness that would require use of general anesthesia (as opposed to sedation) for the MRI.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Drolet, MD, Principal Investigator — Medical College of Wisconsin; Michael Kelly, MD, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Frieden IJ, Reese V, Cohen D. PHACE syndrome. The association of posterior fossa brain malformations, hemangiomas, arterial anomalies, coarctation of the aorta and cardiac defects, and eye abnormalities. Arch Dermatol. 1996 Mar;132(3):307-11. doi: 10.1001/archderm.132.3.307. PMID 8607636
- See also: Children's Hospital of Wisconsin website — http://www.chw.org/display/PPF/DocID/36150/router.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from the Pediatric Dermatology clinic at Children's Hospital of Wisconsin between. Study enrollment period extended from 2008-2009.
Pre-assignment Details: Subjects meeting eligibility criteria including diagnosis and lesional size criteria were enrolled in the study. Subjects who had received topical or intralesional corticosteroids were eligible following a 1 week wash-out period.
Groups:
- Vincristine Treatment Group: Vincristine is a drug that has been used to treat cancers in children (including infants). It has been effective in treating a small number of infants with hemangiomas, most of whom failed previous therapies including steroids. Vincristine must be administered into a vein. Given the encouraging response data and documented safety record, Vincristine is a good choice for a clinical trial treating infants with complicated hemangiomas.
  Vincristine : Vincristine (0.05 mg/kg/dose) will be administered into a vein (PICC line) every week for 12 weeks. If assigned to receive Vincristine, a PICC line will be placed by a doctor who is a specialist in this procedure, an interventional radiologist. This will require sedation and when possible, will be coordinated with sedation for the MRI.
- Oral Steroid Treatment Group: The standard treatment for hemangioma at most centers is oral steroids (Prednisolone). Prednisolone has been used to stop the growth of infantile hemangiomas that are life threatening, that could harm important functions, or are likely to result in severe disfigurement (scarring) without treatment.
  Prednisone : Prednisolone given at 3 mg/kg/day by mouth for 12 week
Period: Overall Study
Arm/Group | Vincristine Treatment Group | Oral Steroid Treatment Group
Started | 4 | 4
Completed | 4 | 1
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vincristine Treatment Group | Oral Steroid Treatment Group | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.18 (0.05) | 0.11 (0.05) | 0.15 (0.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Response of Hemangioma (IH) to Treatment
Description: Response of IH not confined to the dermis will be coded using the following criteria: Progressive disease: >40% increase in volume by MRI, Partial response: >65% reduction in volume by MRI, Complete response: no visual or radiographic evidence of disease, Stable disease: none of the above or <40% increase or <65% decrease in volume by MRI.
  Response of superficial IH will be coded using the following criteria (based on RECIST): Progressive disease: >30% increase in IH size, Partial response: >30% reduction in size, Complete response: no evidence of disease, Stable disease: none of the above.
  Our first 3 patients showed limits to using MRI volume to measure IH size/response to therapy. Unlike other solid tumors, the superficial distribution of some IH made getting volume by MRI difficult, resulting in smaller tumor estimation compared to clinical assessment. Based on these observations, we amended the protocol to report response based on RECIST criteria instead of change in IH volume.
Time Frame: 6 weeks
Population: Per protocol, all participants were analyzed, no matter the treatment arm or treatment success.
Measure: Number; unit: participants
Arm/Group | Vincristine Treatment Group | Oral Steroid Treatment Group
Number analyzed (Participants) | 4 | 3
participants
  Progressive Disease | 0 | 1
  Partial Response | 2 | 0
  Complete Response | 0 | 0
  Stable Disease | 2 | 2

2. Secondary Outcome: Toxicity to Medications
Description: Adverse events were closely monitored and recorded at weekly visits during treatment period and for two years after treatment ceased. Laboratory values were taken every other week during the treatment period.
  Please see Adverse Events module for more details.
Time Frame: Initial visit, 2, 4, 6, 10 and 12 weeks of therapy
Measure: Number; unit: participants
Arm/Group | Vincristine Treatment Group | Oral Steroid Treatment Group
Number analyzed (Participants) | 4 | 4
participants
  Patients with Serious Adverse Events | 0 | 0
  Patients with Other Adverse Events | 3 | 0

ADVERSE EVENTS:
Arm/Group | Vincristine Treatment Group | Oral Steroid Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vincristine Treatment Group (N=4) | Oral Steroid Treatment Group (N=4)
Gastrointestinal: weight loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
obstruction/stenosis of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC (Infections and infestations) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this trial include early termination of enrollment leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No